CLINICAL TRIAL: NCT03231085
Title: Comparison of the Rate of Preoperative Haemoglobin After Administration of Epoetin Alpha Associated With an Oral Medical Supplementation Versus Intravenous Before Surgery of Craniosynostosis at the Child
Acronym: IRON KID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9769; 2016-005065-31 (EudraCT Number)
Record Dates: First submitted 2017-06-27; First posted 2017-07-27 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Craniosynostosis
Keywords: Craniosynostosis; hemoglobin; iron peros; iron intravenous
MeSH Terms: conditions — Craniosynostoses | interventions — ferrous fumarate; Fe(III)-EDTA

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferrous fumarate or ferrostrane (Active Comparator): The oral treatment should begin 21 days before surgery.
  Recommended Dosage ferrous fumarate according to the SPC in force:
  * 5 to 8 kg: 2 cd rases / d or 200mg of ferrous fumarate
  * 8 to 10 kg: 3 cd rases / d or 300mg of ferrous fumarate
  * 10 to 12kg: 4 cd rases / d or 400mg of ferrous fumarate
  Ferrostrane ® (syrup) Laboratory TEOFARMA SRL Either 34mg of iron per teaspoon
  Recommended dosage according to the SPC in force:
  * Infant 5 to 8 kg (about 1 to 6 months): 2 teaspoons a day,
  * Infant from 8 to 12 kg (about 6 to 30 months): 3 teaspoons a day.
  Interventions: Drug: Ferrous fumarate or ferrostrane
- Ferric carboxymaltose (Experimental): The single intravenous treatment the day of the inclusion. Dosage according to: 15mg / kg iron (to dilute in 3 ml / kg of Nacl 0.9% (SSI), to pass in 15 minutes.
  Interventions: Drug: Ferrous fumarate or ferrostrane

INTERVENTIONS:
Drug: Ferrous fumarate or ferrostrane — Young children operated with craniosynostosis and treated with EPO and ferrous fumarate or ferostrane per os or intravenous ferric carboxymaltose.
  Other Names: Intravenous ferric carboxymaltose.

SUMMARY:
Oral iron is commonly used in conjunction with EPO preoperatively for hemorrhagic surgeries in children and especially in the surgery of craniosynostosis. The bioavailability of oral iron is low and compliance with treatment is inconsistent. The aim of this study is to evaluate whether the use of ferric carboxymaltose by injection, which has a much better bioavailability, would make it possible to increase the preoperative hemoglobin level more effectively and thus reduce the risk of perioperative blood transfusion .

DETAILED DESCRIPTION:
Prospective study, randomized in two parallel groups (martial treatment versus venous injection) and stratified by center (Montpellier, Nice, Angers).

The number of subjects required is 100 patients, or 50 per group.

ELIGIBILITY:
Inclusion Criteria:

* Craniosynostosis Surgery
* Age: between 4 and 24 months inclusive
* Weight: less than 12kg
* Hemoglobin: 10 g / dl ≤ Hb 14 ≤ g / dl
* Affiliated patients or beneficiaries of a Social Security scheme
* Signature of the consent of the patient's parents

Exclusion Criteria:

* Generalized infection
* Time for consultation of anesthesia with respect to the date of surgery greater than 5 weeks or less than 22 days.
* Initial biological assessment dating more than 3 months before the consultation of anesthesia
* Parents do not understand French
* BMI greater than 20 kg.m-2
* Contraindications to EPO
* Contraindications to ferric carboxymaltose and to ferrous fumarate

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Variation from reference in hemoglobin rate at the day before surgery | Hemoglobin rate change from reference day (right before treatment) to one day before surgery (from 22 days to 5 weeks maximum)
  Variation of hemoglobin rate between reference value (collected right before the implementation of treatment) and preoperative hemoglobin rate (collected one day before surgery)

SECONDARY OUTCOMES:
Variation from reference in hemoglobin rate at the day before surgery depending on the reference iron status | Reference day (right before treatment) and one day before surgery (from 22 days to 5 weeks maximum)
  Variation of hemoglobin rate between reference value (collected right before the implementation of treatment) and preoperative hemoglobin rate (collected one day before surgery) depending on the reference iron status
Variation from reference in hemoglobin rate at the day before surgery depending on the inflammatory state of patient evaluated by CRP rate before treatment | Reference day (right before treatment) and one day before surgery (from 22 days to 5 weeks maximum)
  Variation of hemoglobin rate between reference value (collected right before the implementation of treatment) and preoperative hemoglobin rate (collected one day before surgery) depending on the CRP rate before treatment
Frequency of EPO treatment discontinuation at the end of 2nd injection | 15 days before surgery
  Number of patient stopping EPO injections at the end of 2nd injection
Variation from reference in iron status at the day before surgery | Reference day (right before treatment) and one day before surgery (from 22 days to 5 weeks maximum)
  Changes in iron status between reference day (right before the implementation of treatment) and preoperative iron status (one day before surgery)
Occurrence of adverse events due to experimental treatments | from treatment administration to end of patient follow-up
  Comparision of adverse event du to experimental treatments (ferric carboxymaltose versus ferrous fumarate)
Compliance of oral iron treatment | At the end of oral iron treatment
  Evaluated by visual analogic scale (0 the minimum to 10 the maximum)
Rate of blood transfusion in perioperative phase and during 3 days following surgery | Perioperative phase and during 3 days following surgery
  Number of transfused patients among all patients
Number of packed red blood cells transfused in perioperative phase and during 3 days following | Perioperative phase and during 3 days following surgery
Volume of packed red blood cells transfused | Perioperative phase and during 3 days following surgery
  Volume in mL/kg
Total perioperative blood loss | Perioperative phase and during 3 days following surgery
  Expressed in red blood cell mass
Cost of oral ferrous fumarate treatment compared to ferric carboxymaltose treatment | At the end of patient folllow-up (6 months after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PIRAT, MD, Principal Investigator — Department d'Anesthésie reanimation Lapeyronie
Locations (2):
- France (2):
  - University Hospital of Angers, Angers
  - University Hospital of Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: No